CLINICAL TRIAL: NCT00731497
Title: Solar Water Disinfections: Randomized Intervention Trial
Brief Title: Solar Water Disinfection Intervention Trial in Bolivia
Acronym: SODIS_Bolivia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Universidad de San Simon (Unknown)
Responsible Party: John M. Colford, Jr., Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AI50087_Register; R01AI050087 (NIH)
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Diarrhea
Keywords: SODIS; Drinking Water; Disinfection; Intervention Trial
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): children in households/villages using Solar Water Disinfection (SODIS) method of disinfecting household drinking water
  Interventions: Device: Solar Water Disinfection (SODIS)
- 2 (No Intervention): children in households/villages where Solar Water Disinfection (SODIS) has not been implemented

INTERVENTIONS:
Device: Solar Water Disinfection (SODIS) — Intervention group has SODIS implemented at the household level as a way to disinfect drinking water
  Other Names: SODIS
  Arms: 1

SUMMARY:
The importance of waterborne gastrointestinal illness throughout the developing world, the existence of a cheap and effective intervention (SODIS), the concurrent limited dissemination program for SODIS, the need for a controlled evaluation of the effectiveness of SODIS under actual field conditions, and the experience of our tri-national collaborative research team in successfully conducting large scale drinking water intervention and observational studies in both the United States and the developing world encourage us to propose the following randomized controlled trial in which our specific aims are to:

* Evaluate the hypothesis that SODIS reduces the incidence of gastrointestinal illness in 660 children under the age of five years in rural Bolivia that are randomly selected from 22 villages ;
* Define, through an extensive microbiologic testing component, the baseline rates of pathogen-specific diarrheal illnesses and the pathogens responsible for the differences in diarrheal illness between active and control groups;
* Document the actual use and acceptance of SODIS by participants in the study;
* Assess the cost-effectiveness of SODIS and the social and economic impact of SODIS at household level;
* Examine through mathematical disease modelling the effects of the presence of multiple transmission pathways within a village on the preventable fraction estimate due to the introduction of SODIS.

DETAILED DESCRIPTION:
More than one third of the population in rural and in peri-urban areas of developing countries has no access to sufficient or clean drinking water free of pathogens. Thus, waterborne gastroenteritis remains a major infrastructural and public health problem particularly, as effective treatment (filtration, chlorination, treatments plants) is often beyond financial means or environmental resources used for water purification (fire-boiling, burning carbon-based fuels) become scarce in those communities. In this context solar disinfection of drinking water is especially appealing using a combination of irradiation by direct sunlight and solar heating to kill the water-borne patho¬gens in contaminated drinking water. To date, the efficacy of the SODIS technology as a home-based, low-cost intervention to provide safe drinking water in low income countries is well established, and a large-scale promotion and dissemination program is under way in seven Latin American countries. The principal objective of this study is to evaluate the effectiveness of home-based solar water disinfection (SODIS) in reducing the burden of gastrointestinal illness in children under 5 years in rural villages participating in a country-wide Bolivian SODIS program. We will conduct a community (cluster)-randomized controlled trial following a cohort of children <5 in each community. Totally, 22 communities will be selected from among those districts designated by the country-program to receive the SODIS intervention. A pair-matched design will be employed where communities are first ranked according to their baseline incidence of diarrheal disease and the intervention then assigned within each of the 11 consecutive pairs of communities randomly to one of them. In each cluster, 30 children (660 in total) will be enrolled and followed up for 12 months. Data on diarrheal illness will be obtained from morbidity diaries kept by mothers and validated through weekly home visits. Stool samples will be collected during the baseline morbidity surveys and at times of a diarrheal episode in a child during follow-up. Water quality monitoring of raw water sources used for drinking water and of water samples after treatment with the SODIS device will be conducted systematically. Mothers of participating children will be interviewed at baseline and during the trial with regard to current water use, behavioral and environmental exposures of their child in the home and within the community. This study will specifically estimate; i.) how much of the efficacy of the SODIS technology established in laboratory experiments and in two tightly control¬led phase-III trials can be retained as effectiveness i.e. under program conditions, ii.) the preventive fraction of all-cause child-diarrhea attributable to SODIS. In addition, pathogen-specific attributable risks of diarrheal illness will be calculated. The project is organised by the University of California, Berkeley, with its substantial experience in water intervention trials in US and it benefits from the tradition of North-South collaboration in public health research of the Swiss Tropical Institute, Basel, Switzerland. It is run jointly with the Universidad Mayor de San Simon which coordinates the Bolivian SODIS program.

ELIGIBILITY:
Inclusion Criteria:

* Consent of Community Leadership
* Permanent residence in village
* Consent of both parents and all other adult household members
* Age 6 months to 5 years

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1163 (Actual)
Dates: Start 2004-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrhea | weekly

SECONDARY OUTCOMES:
analysis of stool | baseline and at diarreal episodes
water quality | systematically

CONTACTS AND LOCATIONS:
Overall Officials: John M Colford, M.D., Ph.D., Principal Investigator — U.C. Berkeley; Daniel Mausezahl, Ph.D., Principal Investigator — Swiss Tropical & Public Health Institute; Andri Christen, Study Director — Bolivia
Locations (2):
- Bolivia (2):
  - Universidad de San Simon, Cochabamba
  - Water and Stool Lab, Totora

REFERENCES:
- [Derived] Christen A, Duran Pacheco G, Hattendorf J, Arnold BF, Cevallos M, Indergand S, Colford JM, Mausezahl D. Factors associated with compliance among users of solar water disinfection in rural Bolivia. BMC Public Health. 2011 Apr 4;11:210. doi: 10.1186/1471-2458-11-210. PMID 21463508
- [Derived] Mausezahl D, Christen A, Pacheco GD, Tellez FA, Iriarte M, Zapata ME, Cevallos M, Hattendorf J, Cattaneo MD, Arnold B, Smith TA, Colford JM Jr. Solar drinking water disinfection (SODIS) to reduce childhood diarrhoea in rural Bolivia: a cluster-randomized, controlled trial. PLoS Med. 2009 Aug;6(8):e1000125. doi: 10.1371/journal.pmed.1000125. Epub 2009 Aug 18. PMID 19688036